CLINICAL TRIAL: NCT05614557
Title: Impact of Silicon-based Formulations on Wound Healing of Laser-induced Microscopic Skin Lesions
Acronym: SPASM11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HealLive; 2022-D0083 (Other: Swissethics)
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention)
- Formulation 1 (Experimental)
  Interventions: Device: Stratacel
- Formulation 2 (Experimental)
  Interventions: Device: Stratamed

INTERVENTIONS:
Device: Stratacel — Silicone-based formulation registered as a European class IIa, TGA (Therapeutic Goods Administration) and FDA listed Class I medical device (wound dressing).
  Arms: Formulation 1
Device: Stratamed — Silicone-based formulation registered as a European class IIa, TGA (Therapeutic Goods Administration) and FDA listed Class I medical device (wound dressing).
  Arms: Formulation 2

SUMMARY:
Delayed wound healing is considered a health problem with devastating consequences for patients, healthcare systems, and societies. Over the past 20 years, many other groups, as well as ourselves, have evaluated various alternatives to improve wound healing. Despite this, the scientific evidence demonstrating the efficacy of recently developed treatments is often limited. Stratacel® and Stratamed® are two gels approved by Swissmedic and the FDA for use in improving wound healing. To this end, the efficacy of these formulations has been visually tested by a physician or by patients. Using the most advanced medical technologies (confocal microscopy and LCOCT), this study aims to investigate the effect of these formulations on the healing of human skin. For this research, a total of 20 volunteers will be included in this study. Volunteers will have up to 7 follow-up appointments over 21 days. Each appointment will last approximately 30 minutes and will be used to perform external measurements of skin healing. All volunteers will use the same formulations (Stratacel® and Stratamed®) with the only difference between volunteers being the anatomical area of application of the formulation. This will be determined by chance. The active participation of the participant is requested for the application of the formulations on the skin twice a day during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers age ≥18 years to 50 years
2. Subjects must be willing and able to participate as required by the protocol.
3. Subjects must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Evidence of any relevant skin or systemic disease (for example diabetes mellitus, cardiovascular disease, hypertension, chronic or acute skin disease) possibly affecting the wound healing of the test site.
2. Any skin alteration (for example tattoo or scar) on the test site.
3. Test sites with terminal hairs
4. Pregnancy or breastfeeding.
5. History of hypertrophic scars or keloid formation or a similar abnormal wound healing.
6. Intake of any drug which in the evaluation of the investigator may interfere with the interpretation of trial results or are known to cause clinically relevant interferences.
7. Body Mass Index (BMI) > 36 kg/m².
8. Have any other condition (including drug abuse, alcohol abuse, or psychiatric disorder) that, in the opinion of the investigator, precludes the patient from following and completing the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of erythema severity via erythema index with and without silicon-based formulations. | 21+-2 days maximum
  Erythema severity is measured using the erythema index (EI). EI will be evaluated by a Mexameter by means of duplicate measurements per skin area in arbitrary units.

SECONDARY OUTCOMES:
Time needed for the scab to fall off | 21+-2 days maximum
  Time needed for the scab to fall off will be evaluated through the study of photo documentation conducted thorough the experiment. To obtain the best possible image of the microscopic treatment zones, a DermLite DL4 dermatoscope will be used. The dermatoscope is a non-invasive device, frequently used in dermatology, which allows a better observation of the skin surface by magnifying it.
Volume of microscopic treatment zones (MTZs) and recovery time | 21+-2 days maximum
  Volume of the MTZs and time to recovery will be evaluated using confocal microscopy. Either by using RCM or LC-OCT (both non-invasive), a minimum of 3 MTZs per region will be evaluated. MTZs will also be evaluated following the classical protocol of biopsy fullowed by H&E staining.

CONTACTS AND LOCATIONS:
Overall Officials: Hans J. Laubauch, Dr. med., Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laubach HJ, Tannous Z, Anderson RR, Manstein D. Skin responses to fractional photothermolysis. Lasers Surg Med. 2006 Feb;38(2):142-9. doi: 10.1002/lsm.20254. PMID 16392146
- [Background] Sandhofer M, Schauer P. The safety, efficacy, and tolerability of a novel silicone gel dressing following dermatological surgery. Skinmed. 2012 Nov-Dec;10(6):S1-7. PMID 23346665
- [Background] Monk EC, Benedetto EA, Benedetto AV. Successful treatment of nonhealing scalp wounds using a silicone gel. Dermatol Surg. 2014 Jan;40(1):76-9. doi: 10.1111/dsu.12366. Epub 2013 Nov 25. No abstract available. PMID 24267314
- [Background] Abdlaty R, Hayward J, Farrell T, Fang Q. Skin erythema and pigmentation: a review of optical assessment techniques. Photodiagnosis Photodyn Ther. 2021 Mar;33:102127. doi: 10.1016/j.pdpdt.2020.102127. Epub 2020 Dec 1. PMID 33276114
- [Background] Garbarino F, Migliorati S, Farnetani F, De Pace B, Ciardo S, Manfredini M, Reggiani Bonetti L, Kaleci S, Chester J, Pellacani G. Nodular skin lesions: correlation of reflectance confocal microscopy and optical coherence tomography features. J Eur Acad Dermatol Venereol. 2020 Jan;34(1):101-111. doi: 10.1111/jdv.15953. Epub 2019 Oct 15. PMID 31520439
- [Derived] Del Rio-Sancho S, Christen-Zaech S, Martinez DA, Punchera J, Guerrier S, Laubach HJ. Line-field confocal optical coherence tomography coupled with artificial intelligence algorithms as tool to investigate wound healing: A prospective, randomized, single-blinded pilot study. J Eur Acad Dermatol Venereol. 2025 Aug;39(8):1481-1488. doi: 10.1111/jdv.20478. Epub 2024 Dec 17. PMID 39688344
- [Derived] Del Rio-Sancho S, Christen-Zaech S, Alvarez Martinez D, Punchera J, Merat R, Laubach HJ. Comparing Line-Field Confocal Optical Coherence Tomography and Reflectance Confocal Microscopy on the In Vivo Healing Process of Lesions Induced by Fractional Photothermolysis. Lasers Surg Med. 2025 Jan;57(1):121-129. doi: 10.1002/lsm.23841. Epub 2024 Sep 8. PMID 39245876